CLINICAL TRIAL: NCT04583176
Title: Measurement of Physical Activity in the First Days After Thoracic Surgery
Acronym: Marchez
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_0046
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Disease
Keywords: ActiGraph GT3X; Physical activity
MeSH Terms: conditions — Lung Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective measurement of physical activity has several advantages compared to declarative measures: exemption from memory bias and desirability bias, more precise evaluation, taken into account activities of low intensity, measurement of physical activity and sedentariness profiles (number and duration of periods of activity, number of breaks in sedentary lifestyles).

The aim of this study is to assess the early postoperative mobility of patients who have undergone pulmonary excision by thoracoscopy or robot surgery using ActiGraph GT3X accelerometer. This assessment will serve as a reference element for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Having to undergo pulmonary excision by thoracoscopy or robotic surgery
* Accepting to wear a belt fitted with an ActiGraph GT3X accelerometer for a maximum of 5 days post surgery
* Affiliated to a Health Insurance plan
* Having given an oral non-opposition

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient unable to move independently (paraplegic, etc.)
* Patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having to undergo pulmonary excision by thoracoscopy or robotic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Measurement of postoperative mobility during the first postoperative days | Day 5
  Number of steps

SECONDARY OUTCOMES:
Volume of physical activity assessed by accelerometry during the first postoperative days | Day 5
  Total activity counts per day
Overall intensity of physical activity assessed by accelerometry during the first postoperative days | Day 5
  Steps and counts per hour and per minute
Duration and intensity of physical activity assessed by accelerometry during the first postoperative days | Day 5
  Time in physical activity of different intensities
Sedentary time assessed by accelerometry during the first postoperative days | Day 5
  Total sedentary time
Best natural effort assessed by accelerometry during the first postoperative days | Day 5
  Peak cadence
Patterns of physical activity assessed by accelerometry during the first postoperative days | Day 5
  Number and mean duration of bouts of physical activity
Patterns of sedentary behavior assessed by accelerometry during the first postoperative days | Day 5
  Number and mean duration of bouts of sedentary behavior
Physiotherapists' evaluation during the first post-operative days | Day 5
  Daily activity assessment after thoracic surgery Questionnaire
Postoperative analgesia | Day 5
  Daily activity assessment after thoracic surgery Questionnaire
Assessement of patient acceptability for wearing the ActiGraph GT3X | Day 5
  Digital assessment scale
Postoperative complications | Day 5
  Morbidity and Mortality after Thoracic Surgery Classification

CONTACTS AND LOCATIONS:
Overall Officials: Julien FESSLER, MD, Principal Investigator — Foch Hospital; Marc FISCHLER, PhD, Study Chair — Foch Hospital
Locations (1):
- Hôpital Foch, Suresnes, France